CLINICAL TRIAL: NCT07201987
Title: Intraoperative Placement of Vancomycin-impregnated Calcium Sulfate Beads Conjugated With Analgesics to Improve Spine Surgery Outcomes
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ganesh M. Shankar (Other)
Responsible Party: Sponsor-Investigator, Ganesh M. Shankar, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025p001993
Record Dates: First submitted 2025-09-08; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Spine Surgery; Postoperative Pain Management
Keywords: Spine surgery; Postoperative pain management; Calcium sulfate beads; Vancomycin; Analgesics; Hospital length of stay
MeSH Terms: interventions — Vancomycin; Morphine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vancomycin-impregnated calcium sulfate beads with morphine and bupivacaine (Experimental): Patients will receive intraoperative placement of vancomycin-impregnated calcium sulfate beads conjugated with morphine and bupivacaine for pain control, in addition to standard perioperative care.
  Interventions: Drug: Vancomycin (local, via calcium sulfate beads); Drug: Morphine (local, via calcium sulfate beads); Drug: Bupivacaine (local, via calcium sulfate beads)
- Vancomycin-impregnated calcium sulfate beads (standard-of-care) (Active Comparator): Patients will receive intraoperative placement of vancomycin-impregnated calcium sulfate beads for surgical site infection prophylaxis, without added analgesics.
  Interventions: Drug: Vancomycin (local, via calcium sulfate beads)

INTERVENTIONS:
Drug: Vancomycin (local, via calcium sulfate beads) — Patients undergoing spine surgery will receive intraoperative placement of calcium sulfate beads impregnated with vancomycin. The beads are intended to provide local infection prophylaxis.
Drug: Morphine (local, via calcium sulfate beads) — Patients undergoing spine surgery in the experimental arm will receive intraoperative placement of calcium sulfate beads impregnated with morphine. The beads are intended to provide sustained local analgesia.
  Arms: Vancomycin-impregnated calcium sulfate beads with morphine and bupivacaine
Drug: Bupivacaine (local, via calcium sulfate beads) — Patients undergoing spine surgery in the experimental arm will receive intraoperative placement of calcium sulfate beads impregnated with bupivacaine. The beads are intended to provide sustained local analgesia.
  Arms: Vancomycin-impregnated calcium sulfate beads with morphine and bupivacaine

SUMMARY:
The goal of this clinical trial is to learn if using calcium sulfate beads that contain vancomycin (an antibiotic) and pain-relieving medicines during spine surgery can improve recovery compared to standard care with intravenous (IV) morphine and local pain medicines.

Researchers want to know if the sustained release formulation of morphine from these calcium sulfate beads affect:

* Postoperative length of stay
* Postoperative pain scores
* Postoperative narcotic analgesic requirements

All participants in this study will already be scheduled to have spine surgery as part of their regular medical care. During surgery, participants will be assigned to receive either intraoperative placement of calcium sulfate beads with vancomycin alone or vancomycin with morphine and bupivacaine. All patients will still have access to standard of care with IV and PO pain regimens. Participants will then be followed after surgery to measure their pain, recovery, and medication use.

Participation is voluntary, and choosing not to join will not affect a person's medical care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to understand and provide consent in English
* Undergoing elective lumbar spinal decompression and fusion surgery at one or two levels

Exclusion Criteria:

* History of allergy or hypersensitivity to morphine, bupivacaine, or calcium sulfate.
* Active systemic or localized infection at the surgical site.
* History of chronic opioid dependence or opioid use disorder (as it may confound pain assessment).
* Patients with severe renal or hepatic impairment (due to altered metabolism of analgesics and risk of complications from analgesic side effects).
* Pregnant or breastfeeding individuals.
* Filling of defects that are intrinsic to the stability of the bony structure
* Severe vascular or neurological disease
* Uncontrolled diabetes
* Severe degenerative bone disease
* Hypercalcemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Total Postoperative Analgesic Consumption in Morphine Milligram Equivalents (MME) | From end of surgery through 8 weeks post-surgery.
  Cumulative dose of opioids and non-opioid analgesics used postoperatively, converted to morphine milligram equivalents.
Change from Baseline in Postoperative Pain Intensity as Measured by PROMIS Pain Intensity Short Form 3a | Baseline (pre-surgery), 24-48 hours, 2-3 weeks, and 8 weeks post-surgery.
  Average change in self-reported pain intensity using the PROMIS Pain Intensity Short Form 3a, scored on a 0-10 scale (0 = no pain, 10 = worst possible pain).
Length of Hospital Stay | From the day of surgery until hospital discharge (typically 2-7 days postoperatively)
  Number of days from surgery to hospital discharge.
Change from Baseline in Functional Status as Measured by PROMIS Physical Function Short Form 10a | Baseline (pre-surgery), 2-3 weeks, and 8 weeks post-surgery.
  Change in physical function as reported by participants using the PROMIS Physical Function Short Form 10a. Scores are reported as T-scores (mean = 50, SD = 10); higher scores indicate better function.
Change from Baseline in Functional Status as Measured by Oswestry Disability Index (ODI) | Baseline (pre-surgery), 2-3 weeks, and 8 weeks post-surgery.
  Change in disability as reported by participants using the Oswestry Disability Index (ODI). Scores range from 0 to 100; higher scores indicate greater disability.

SECONDARY OUTCOMES:
Incidence of Surgical Site Infections | Within 8 weeks post-surgery.
  Number of participants with a postoperative surgical site infection, defined by CDC criteria.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcome results (including demographics, pain scores, analgesic consumption, hospital length of stay, functional outcomes, and adverse event data) will be shared. No data containing direct identifiers will be provided.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD and supporting documents will be made available beginning 6 months after publication of the primary study results and will remain available for 5 years.
Access Criteria: Access will be granted to qualified researchers affiliated with academic or healthcare institutions who provide a methodologically sound proposal for secondary analyses related to spine surgery outcomes, pain management, or infection prevention. Proposals will be reviewed by the Principal Investigator and research team. Upon approval, data will be shared via a secure, HIPAA-compliant institutional data-sharing platform. Requests should be directed to Ganesh Shankar (gshankar@mgh.harvard.edu).